CLINICAL TRIAL: NCT04240535
Title: A Single Center, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of OnabotulinumtoxinA to the Depressor Anguli Oris
Brief Title: Evaluation of the Safety and Efficacy of OnabotulinumtoxinA to the Depressor Anguli Oris
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amir Moradi MD, MBA (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Amir Moradi MD, MBA, Principal Investigator, Moradi MD
Organization: Moradi MD (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMD103
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Aging
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active- onabotulinumtoxinA (Experimental): BOTOX Cosmetic (onabotulinumtoxinA) for injection, is a sterile, vacuum-dried purified botulinum toxin type A, produced from fermentation of Hall strain Clostridium botulinum type A intended for intramuscular use. It is purified from the culture solution by dialysis and a series of acid precipitations to a complex consisting of the neurotoxin, and several accessory proteins. The complex is dissolved in sterile sodium chloride solution containing Albumin Human and is sterile filtered (0.2 microns) prior to filling and vacuum-drying.
  Interventions: Drug: OnabotulinumtoxinA 50 UNT [Botox Cosmetic]
- Placebo-Bacteriostatic 0.9% Sodium Chloride (Placebo Comparator): Placebo subjects will have injections in the same manner, but will be injected with Bacteriostatic 0.9% Sodium Chloride.
  Interventions: Drug: OnabotulinumtoxinA 50 UNT [Botox Cosmetic]

INTERVENTIONS:
Drug: OnabotulinumtoxinA 50 UNT [Botox Cosmetic] — Injections to the Depressor Anguli Oris
  Other Names: Botox Cosmetic

SUMMARY:
Single Center, Double Blind, Placebo- Controlled Study of 20 subjects with 10 active drug/10 placebo

Standardized baseline/pre-treatments and follow-up images will be taken.

Subjects will receive injection of either study drug or placebo to the Depressor Anguli Oris. Follow ups will occur at 2 weeks, 4 weeks, and 12 weeks.

DETAILED DESCRIPTION:
1. This study is a prospective single-center, clinical trial to be conducted at one clinical site. Up to 20 subjects will be enrolled and treated (total enrollment may be more than 20 due to screen failures) if they meet the inclusion/exclusion criteria and provide written informed consent.
2. Duration of Study The duration from when the study opens to enrollment until completion of data analysis is anticipated to be six months
3. Study Endpoints 3.1 Primary Endpoint: One grade improvement on Depressor Anguli Oris Scale as assessed by the Principal Investigator

Depressor Anguli Oris Scale

0-None Slight or no muscle contraction

1. Mild Mild contraction with mild pull down of corner of the mouth
2. Moderate Moderate muscle contraction and moderate pull down of corner of mouth
3. Severe Severe Muscle contraction with sever pull down of corner of the mouth

3.2 Secondary Endpoints

The secondary endpoints of this clinical trial include:

1. The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a Global Aesthetic Improvement Scale (Investigator Global Aesthetic Improvement Scale) assessing overall aesthetic improvement at 2 weeks, 6 weeks, and 12 weeks after the treatment visit.
2. The subjects will complete the Global Aesthetic Improvement Scale (Subject Global Aesthetic Improvement Scale) assessing overall aesthetic improvement at 2 weeks, 6 weeks, and 12 weeks after the treatment visit.
3. The subject will complete a Patient Satisfaction Questionnaire at 2 weeks, 6 weeks, and 12 weeks after the treatment visit.
4. Analysis of photography to provide data on change in facial muscle contraction

4. Outcome Measures 4.1 The Global Aesthetic Improvement Scale is a 5-point scale that rates global aesthetic improvement from the pretreatment appearance. The ratings are worse, no change, improved, much improved, and very much improved. In this study both live observation and photo review are utilized by the physician or a qualified, delegated clinician and subject in order to assign a score. The Investigator Global Aesthetic Improvement Scale must be performed by the principal investigator, sub-investigator or qualified clinician delegated by the principal investigator.

4.2 Subject Satisfaction Questionnaire Part A (Baseline Only Visit)

1. How satisfied are you with your appearance?

   - Very satisfied
   * Satisfied
   * Slightly satisfied
   * Neither satisfied or dissatisfied
   * Dissatisfied
2. Which statement do you agree with?

   * I look younger than my age
   * I look my current age
   * I look older than my age

Subject Satisfaction Questionnaire Part B

1. How satisfied are you with your appearance?

   - Very satisfied

   - Satisfied
   * Slightly satisfied
   * Neither satisfied or dissatisfied
   * Dissatisfied
2. Which statement do you agree with?

   - I look younger than my age

   - I look my current age

   - I look older than my age
3. Do you notice any improvement in how your skin looks in the area that was treated?

   - Yes

   - No
4. How would you characterize your satisfaction with the treatment?

   - Very satisfied

   - Satisfied
   * Slightly satisfied
   * Neither satisfied or dissatisfied
   * Dissatisfied
5. Would you recommend the treatment to your friends and family members? (check one)

   * Yes
   * No

5. Subject enrollment 5.1 Participant Inclusion Criteria The study population will consist of males and females aged 18 years and older who have chosen to participate in this clinical trial as evidenced by execution of the informed consent document. 10 subjects will receive treatment and 10 subjects will receive placebo.

5.1.1 Informed Consent Written informed consent will be obtained from all subjects (or their guardians or legal representatives) before any study-related procedures, including any pre-treatment screening procedures, are performed. Investigators, or delegated study personnel, may discuss the availability of the study and the possibility for entry with a potential subject without first obtaining consent. Informed consent must be obtained and documented prior to initiation of any procedures that are performed solely for the purpose of determining eligibility for research.

Investigators have ethical and legal responsibilities to ensure that the protocol is clearly explained to each subject considered for enrollment in the study. Compliance with this requirement should be documented on a written Informed Consent Form approved by the reviewing Institutional Review Board. Each Informed Consent Form will include the elements required by Food and Drug Administration regulations in 21 Code of Federal Regulations Part 50.

The Institutional Review Board approved Informed Consent Form will be signed by the study personnel obtaining consent. The subject will be given a copy of the signed Informed Consent Form. The investigative site will keep the original on file.

6. Study Drug BOTOX Cosmetic (onabotulinumtoxinA) for injection, is a sterile, vacuum-dried purified botulinum toxin type A, produced from fermentation of Hall strain Clostridium botulinum type A intended for intramuscular use. It is purified from the culture solution by dialysis and a series of acid precipitations to a complex consisting of the neurotoxin, and several accessory proteins. The complex is dissolved in sterile sodium chloride solution containing Albumin Human and is sterile filtered (0.2 microns) prior to filling and vacuum-drying.

The primary release procedure for BOTOX Cosmetic uses a cell-based potency assay to determine the potency relative to a reference standard. The assay is specific to Allergan's products BOTOX and BOTOX Cosmetic. One Unit of BOTOX Cosmetic corresponds to calculated median intraperitoneal lethal dose in mice. Due to specific details of this assay such as the vehicle, dilution scheme and laboratory protocols, Units of biological activity of BOTOX Cosmetic cannot be compared to nor converted into Units of any other botulinum toxin or any toxin assessed with any other specific assay method. The specific activity of BOTOX Cosmetic is approximately 20 Units/nanogram of neurotoxin complex.

Each vial of BOTOX Cosmetic contains either 50 Units of Clostridium botulinum type A neurotoxin complex, 0.25 mg of Albumin Human, and 0.45 mg of sodium chloride; or 100 Units of Clostridium botulinum type A neurotoxin complex, 0.5 mg of Albumin Human, and 0.9 mg of sodium chloride in a sterile, vacuum-dried form without a preservative.

7. Study Procedures and Schedule 7.1 Study Images Standardized baseline and follow-up images will be taken. To ensure consistent, reproducible study photos from baseline photographs to the follow-up photographs, Moradi MD's study specific photography guidelines and procedures should be followed.

8 Study Schedule Visit 1-Screening, Baseline & Treatment

* Obtain informed consent of potential participant verified by signature on study informed consent form.
* Verify all preliminary/screening inclusion/exclusion criteria are met.
* Document medical history.
* Investigator skin assessment
* Obtain pregnancy screen (if applicable).
* Safety assessments
* Focused physical examination
* Subject satisfaction questionnaire part A
* Perform baseline photography.
* Document concurrent medications.
* Obtain demographics.
* Perform study treatment.
* Assess for expected treatment effects and adverse events

Visit 2- 2 week follow up visit (+/- 4 days)

* Obtain images.
* Assess for expected treatment effects and adverse events
* Obtain aesthetic improvement scores
* Obtain patient satisfaction questionnaire
* Obtain Depressor Anguli Oris Scale Score by Principal Investigator
* Focused physical examination
* Subject satisfaction questionnaire part B
* Safety Assessments

Visit 3-4 week follow up visit (+/-7 days)

* Obtain images.
* Assess for expected treatment effects and adverse events
* Obtain aesthetic improvement scores
* Obtain patient satisfaction questionnaire
* Obtain Depressor Anguli Oris Scale Score by Principal Investigator
* Focused physical examination
* Subject satisfaction questionnaire part B
* Safety Assessments

Visit 4- 12 week follow up visit (+/-7 days)

• Obtain images.

* Assess for expected treatment effects and adverse events
* Obtain aesthetic improvement scores
* Obtain patient satisfaction questionnaire
* Obtain Depressor Anguli Oris Scale Score by Principal Investigator
* Focused physical examination
* Subject satisfaction questionnaire part B
* Safety Assessments

  9. Unscheduled Visit Any unscheduled visit or examine should be documented in the subject's medical record and adverse event form (if applicable) stating the reason for the visit and any actions taken.

  10. Study Treatments This study involves a treatment of either onabonulinumtoxin A or a placebo to be injected in the Depressor Anguli Oris after obtaining informed consent, screening for inclusion/exclusion, complying with standardized photography requirements, and completing pregnancy tests, if applicable.

  11. Pre-Treatment Medications For this protocol, pre-treatment medication will be at the investigator's discretion and will be documented accordingly.

  12. Subject Preparation for Treatment The investigator, sub-investigator, or delegated clinician will first identify the skin areas to which treatment is to be performed. Treatment records for all regions will be maintained in accordance with this protocol. Skin in target treatment area should be cleansed with mild cleaner. No lotion, make-up, perfume, powder, or oil should be present on the area to be treated.

  13. Treatment All study treatments will be performed by the Investigator. For the study treatment 4.5 units of Botox Cosmetic will be injected per side in three injection points. Each injection point is 1.5 units of Botox for a total of six injection point, with a total of nine units. First injection is just below and lateral to the oral commisure where the skin dimples upon activation of the Depressor Anguli Oris. The second injection is between 1st and 3rd injection points along the same oblique line. The third injection is more laterally and at the mid distance from oral commisure to Jawline, along the line of Depressor Anguli Oris

Placebo subjects will have injections in the same manner, but will be injected with Bacteriostatic 0.9% Sodium Chloride.

The subjects will be monitored during the treatment for Adverse Events.

14. Concomitant Medications All concomitant prescription, non-prescription and over-the-counter medications taken during study participation will be recorded on the appropriate study-specific data form. For this protocol, a prescription medication is defined as a medication that can be prescribed only by a properly authorized/licensed clinician.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
2. Male or non-pregnant, non-breastfeeding females
3. Age ranging between 18-65
4. Subject seeking augmentation therapy of the depressor anguli oris.
5. Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the horizontal line from the sub nasal for the duration of the study. (e.g. laser or chemical peels, skin resurfacing, microdermabrasion, etc.)
6. If the subject is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test at the screening/enrollment visit and prior to treatment.

   Acceptable forms of effective birth control include:

   Barrier methods of contraception: Condom or Occlusive cap
   * (diaphragm or cervical caps) with spermicidal foam/gel/film/cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or Injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to baseline and agrees to continue for the duration of the study or use acceptable form of birth control). Negative urine pregnancy test at screening.
7. Subjects willing to provide written consent for use of photography -

Exclusion Criteria:

1. History of other facial treatment/procedure in the previous 6 months below the level of the horizontal line from sub nasal that, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessments or exposes the subject to undue risk by study participation.
2. Presence of any disease or lesions near or on the area to be treated:

   * Inflammation, active or chronic infection (e.g., in mouth, dentals, head and neck region);
   * Facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes simplex or herpes zoster;
   * Scars or deformities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
One grade improvement on Depressor Anguli Oris Scale | 2 weeks Post Treatment
  The scale will be used to measure if the subject has had any grade improvement in the treated area since baseline. Scale measures the severity of the depressor Anguli Oris from a 0-none-3 Severe as explained in the Detailed description section 3

SECONDARY OUTCOMES:
Improvement on Investigator Global Aesthetic Improvement Scale | 2 weeks Post Treatment
  The Global Aesthetic Improvement Scale is a 5-point scale that rates global aesthetic improvement from the pretreatment appearance.Global Aesthetic Scale is defined in Detailed Description Section 4
Improvement on Subject Global Aesthetic Scale | 2 weeks Post Treatment
  The Global Aesthetic Improvement Scale is a 5-point scale that rates global aesthetic improvement from the pretreatment appearance.this one will be fore the subject. The Global Aesthetic Scale is defined in Detailed Description Section 4.
Patient Satisfaction Questionnaire | 2 weeks Post Treatment
  This questionnaire will be used to measure the level of satisfication if any since the subject was treated in the Depressor Anguli Oris. A detailed list of the questions is in the Detailed Description Section 4
Photographic Analysis | 2 weeks Post Treatment
  Analysis of photography to provide or confirm change in facial muscle contraction. Subjects will use the images help score when using the Using the subject Global aesthetic Scale.
Safety Assessments such as Focused Physical & adverse event, or expected treatment effects | 12 weeks Post Treatment
  Number of participants with treatment- related adverse events as assessed by Principal Investigator will occur at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moradi, MD, MBA, Principal Investigator — Moradi MD
Locations (1):
- Moradi MD, Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moradi A, Khalifian S, Alghoul MS, Poehler J. A Novel 3-Point Injection Technique for OnabotulinumtoxinA in the Upper Depressor Anguli Oris. Dermatol Surg. 2023 Mar 1;49(3):259-265. doi: 10.1097/DSS.0000000000003695. Epub 2023 Feb 10. PMID 36763899